CLINICAL TRIAL: NCT04936152
Title: Effects of Mirror Therapy Application of Tablet pc on Acute Bell's Palsy.
Brief Title: Mirror Therapy on PC in Acute Bell's Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00658 Ameemah Talib
Record Dates: First submitted 2020-12-21; First posted 2021-06-23 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; mime therapy; mirror therapy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mime therapy using tablet PC mirror application (Active Comparator): these individuals will receive mime therapy using tablet PC mirror application
  Interventions: Other: mime therapy using tablet PC mirror application
- the control intervention including the mime therapy (Experimental): these individuals will receive the control intervention including the mime therapy).
  Interventions: Other: the control intervention including the mime therapy

INTERVENTIONS:
Other: mime therapy using tablet PC mirror application — After the baseline assessment, The patient in the experimental group will receive mirror therapy and mime therapy.
  Exercises time period is 30 min/session
  Mime Therapy Using Tablet PC:
  Mirror therapy using tablet PC mirror application We will use a tablet PC mirror application that can convert images from right to left. In the mirror group, the mirror application was used during the exercise. Patients watched the tablet PC screen. The mirror application converts the image from right to left.
  • Mime therapy include Mime therapy will consists of auto massage- effleurage and kneading for 10 to 15minutes on both the sides of the face, stretching exercises of the muscles of the affected side followed by facilitation, specific low intensity exercises to co-ordinate both the halves of the face, active assisted exercises for affected side of the face, exercises of mouth and eye with simultaneous inhibition of synkinesis if present.
  Arms: mime therapy using tablet PC mirror application
Other: the control intervention including the mime therapy — After the baseline assessment, The patient in the experimental group will receive mime therapy Mime therapy include Mime therapy will consists of auto massage- effleurage and kneading for 10 to 15minutes on both the sides of the face, stretching exercises of the muscles of the affected side followed by facilitation, specific low intensity exercises to co-ordinate both the halves of the face, active assisted exercises for affected side of the face, exercises of mouth and eye with simultaneous inhibition of synkinesis if present.
  Arms: the control intervention including the mime therapy

SUMMARY:
The objective of this study is to compare the effects of mime therapy using mirror therapy application of tablet PC vs mime therapy on acute bell's palsy. Study Design was Randomized control trial with Sample Size was 22. Sampling Technique was Purposive sampling. Randomization was done through a sealed envelope method. Study Setting included Physiotherapy department of DHQ Teaching Hospital, Mirpur Azad Kashmir. Inclusion criteria were Age between 30-60year, Both male & female and Acute bell's palsy ( 2-3 weeks). Exclusion criteria were Individuals with the other neurological deficits, Visual impairment, History of facial palsy of central type, Surgical intervention for ear and facial nerve palsy and Non-co-operative patients. tools used for assessment was Sunnybrook Facial Grading system scale, House-Brackmann Facial Grading System and Patients Global Impression of Change. Individuals who met the inclusion criteria were included in this study. All participants went through randomization and divided into two groups Experimental group 1 (these individuals will receive mime therapy using tablet PC mirror application)and Experimental group 2 (these individuals will receive the control intervention including the mime therapy). Pre-intervention assessment is made for both groups. Then intervention will apply to both groups. Estimated time of treatment protocol will be 30 minutes session, 4 times/week for 4 weeks in the hospital setting. Subjects will be evaluated at baseline, then 2nd week and 4th-week assessment will be the final. All statistical analyses were performed through SPSS 21. Normality of data was assessed and after checking normality parametric or non-parametric test was applied accordingly.

.

DETAILED DESCRIPTION:
Damage or dysfunction of the facial nerve can result in paralysis, abnormal muscle tone, abnormal movement patterns, eye irritations, and decreased facial expression. Medical conditions that can typically result in facial nerve dysfunction are Bell's palsy, herpesvirus, temporal bone fracture, facial or head trauma, acoustic neuroma excision, facial nerve schwannoma, vascular damage, and neoplasms. The facial nerve sustains impairment more often than any other nerve in the body. The term Bells' Palsy is defined as an idiopathic, acute and unilateral paresis or paralysis of the face which may be partial or complete occurring with equal frequencies on right and left sides of the face. The major cause of Bell's Palsy is idiopathic, accounting for 50% of all cases. Other few suggested causes are exposure to cold, middle ear infections, dental and ENT surgeries and traumatic. The problems faced in the acute phase of Bell's palsy include difficulty in closing the affected side-eye, facial deviation to the unaffected side, difficulty in drinking, eating and speaking along with psychological problems and facial appearance is the main concern in any phase of Bell's palsy. Complete recovery of facial function in Bell's palsy occurs in 70% of people within three months (Peitersen 1994) with about 30% of people continuing to suffer facial asymmetry at rest and during movement, as well as synkinesis. Treatment of Bell's palsy is controversial due to the lack of large, randomized, controlled, prospective studies. There are indications that steroids or antiviral agents are beneficial but also studies, which show no beneficial effect. Additional measures include eye protection, physiotherapy, acupuncture, botulinum toxin, or possibly surgery. A Cochrane review done by in February 2011 has concluded that there is only very low-quality evidence that facial exercise reduces sequel in acute cases. A study done in 2009 has concluded that massage done in mime therapy has shown to create new growth and increase the production of collagen and connective tissue in facial muscles and restore facial muscle action. A study done on mime therapy efficacy in patients with long term facial nerve paresis shows that mime therapy improves facial symmetry.A study of 2014 observed the half-mirror biofeedback exercise in combination with three botulinum toxin after facial paralysis. Half-mirror biofeedback rehabilitation designed for facial sequelae shows good results in combination with botulinum toxin therapy. This facial rehabilitation strategy, consisting of three injections of botulinum toxin and half-mirror biofeedback exercises, proceeds over the course of 2 years and offers a long-lasting cure for facial synkinesis and facial symmetry as well as improved facial aesthetics. A study in 2011 on facial biofeedback rehabilitation with a mirror after administration of a single dose of botulinum A toxin on facial synkinesis was examined in patients with chronic facial palsy concluded that Facial biofeedback rehabilitation with a mirror after administration of a single dose of botulinum A toxin can be a long-lasting treatment of established facial synkinesis. A study of, 2013 Mime therapy improves facial symmetry and functions more than conventional therapy and home exercises in people with acute Bell's Palsy. No difference was found between conventional therapy and home exercise program. A study in, 2016 investigate the effects of mirror therapy using a tablet PC for post-stroke central facial paresis. A prospective, randomized controlled study was performed. Twenty-one post-stroke patients were enrolled. All patients performed 15 minutes of orofacial exercise twice daily for 14 days concluded that mirror therapy using a tablet PC might be an effective tool for treating central facial paresis after stroke. The past research records are evident that therapists have worked with mime therapy and mirror therapy. The two protocols have not been complimented for rehabilitation. So the aim of this study is to observe and determine the combined effect of these two treatment protocols to get the results and improve the facial symmetry in acute bell's palsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute bell's palsy ( 2-3 weeks)

Exclusion Criteria:

* Individuals with the other neurological deficits
* Visual impairment
* History of facial palsy of central type
* Surgical intervention for ear and facial nerve palsy.
* Non co-operative patients.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Sunnybrook Facial Grading system scale | 4 weeks
  The Sunnybrook facial grading scale is a regionally weighted system that includes evaluation of resting symmetry, degree of voluntary movements and synkinesis to form a composite score from 0 to 100, where 0 is complete paralysis and 100 normal facial functions.
  The tool will be used for assessment.

OTHER OUTCOMES:
House-Brackmann Facial Grading System | 4 weeks
  The House-Brackmann Facial Nerve Grading System is widely used to characterize the degree of facial paralysis. In this scale, grade I is assigned to normal function, and grade VI represents complete paralysis. Intermediate grades vary according to function at rest and with effort.
  The tool will be used for assessment
Patients Global Impression of Change | 4 weeks
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. PGIC remains a clinically relevant tool to assess perceived impact of disease management.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronin GW, Steenerson RL. The effectiveness of neuromuscular facial retraining combined with electromyography in facial paralysis rehabilitation. Otolaryngol Head Neck Surg. 2003 Apr;128(4):534-8. doi: 10.1016/S0194-59980300005-6. PMID 12707657
- [Background] Santos MA, Caiaffa Filho HH, Vianna MF, Almeida AG, Lazarini PR. Varicella zoster virus in Bell's palsy: a prospective study. Braz J Otorhinolaryngol. 2010 May-Jun;76(3):370-3. doi: 10.1590/S1808-86942010000300016. PMID 20658018
- [Background] Devriese PP. Rehabilitation of facial expression ("mime therapy"). Eur Arch Otorhinolaryngol. 1994 Dec:S42-3. No abstract available. PMID 10774308
- [Background] Baugh RF, Basura GJ, Ishii LE, Schwartz SR, Drumheller CM, Burkholder R, Deckard NA, Dawson C, Driscoll C, Gillespie MB, Gurgel RK, Halperin J, Khalid AN, Kumar KA, Micco A, Munsell D, Rosenbaum S, Vaughan W. Clinical practice guideline: Bell's palsy. Otolaryngol Head Neck Surg. 2013 Nov;149(3 Suppl):S1-27. doi: 10.1177/0194599813505967. PMID 24189771
- [Background] Beurskens CH, Heymans PG. Mime therapy improves facial symmetry in people with long-term facial nerve paresis: a randomised controlled trial. Aust J Physiother. 2006;52(3):177-83. doi: 10.1016/s0004-9514(06)70026-5. PMID 16942452
- [Background] Finsterer J. Management of peripheral facial nerve palsy. Eur Arch Otorhinolaryngol. 2008 Jul;265(7):743-52. doi: 10.1007/s00405-008-0646-4. Epub 2008 Mar 27. PMID 18368417
- [Background] Teixeira LJ, Soares BG, Vieira VP, Prado GF. Physical therapy for Bell s palsy (idiopathic facial paralysis). Cochrane Database Syst Rev. 2008 Jul 16;(3):CD006283. doi: 10.1002/14651858.CD006283.pub2. PMID 18646144
- [Background] Lee JM, Choi KH, Lim BW, Kim MW, Kim J. Half-mirror biofeedback exercise in combination with three botulinum toxin A injections for long-lasting treatment of facial sequelae after facial paralysis. J Plast Reconstr Aesthet Surg. 2015 Jan;68(1):71-8. doi: 10.1016/j.bjps.2014.08.067. Epub 2014 Sep 18. PMID 25444667
- [Background] Azuma T, Nakamura K, Takahashi M, Ohyama S, Toda N, Iwasaki H, Kalubi B, Takeda N. Mirror biofeedback rehabilitation after administration of single-dose botulinum toxin for treatment of facial synkinesis. Otolaryngol Head Neck Surg. 2012 Jan;146(1):40-5. doi: 10.1177/0194599811424125. Epub 2011 Sep 30. PMID 21965443
- [Background] Kang JA, Chun MH, Choi SJ, Chang MC, Yi YG. Effects of Mirror Therapy Using a Tablet PC on Central Facial Paresis in Stroke Patients. Ann Rehabil Med. 2017 Jun;41(3):347-353. doi: 10.5535/arm.2017.41.3.347. Epub 2017 Jun 29. PMID 28758071
- [Background] Neely JG, Cherian NG, Dickerson CB, Nedzelski JM. Sunnybrook facial grading system: reliability and criteria for grading. Laryngoscope. 2010 May;120(5):1038-45. doi: 10.1002/lary.20868. PMID 20422701
- [Background] Reitzen SD, Babb JS, Lalwani AK. Significance and reliability of the House-Brackmann grading system for regional facial nerve function. Otolaryngol Head Neck Surg. 2009 Feb;140(2):154-8. doi: 10.1016/j.otohns.2008.11.021. PMID 19201280